CLINICAL TRIAL: NCT05810688
Title: Aspiration Pneumonia is High Morbidity and Mortality Rate. Nasogastric Tube Insertion is an Emergency Medical Treatment. The Results of the Successful Strategy for Removing Senior Aspiration Pneumonia Patient's Nasogastric Tubes.
Brief Title: Eating Rehabilitation Training for Timely Removal of Nasogastric Tube in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD professer, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TPEVGH 2023-01-005AC
Record Dates: First submitted 2023-03-19; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Aspiration Pneumonia
Keywords: elderly; Aspiration Pneumonia; eating rehabilitation training; removal of nasogastric tube
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating rehabilitation training group (Experimental): The intervention group will receive eating rehabilitation training, including oral care, saliva gland massage, oral exercise, feeding strategy, and swallowing skill education
  Interventions: Other: eating rehabilitation training
- Control group (No Intervention): The control group will receive only usual care.

INTERVENTIONS:
Other: eating rehabilitation training — The experimental group will receive eating rehabilitation training, including oral care, saliva gland massage, oral exercise, feeding strategy, and swallowing skill education.
  Arms: Eating rehabilitation training group

SUMMARY:
Aspiration pneumonia is a common complication in senior patients with high morbidity and mortality rate. The decline of physical function among elders can easily lead to swallowing disorders, and nasogastric (NG) tube insertion is an emergency medical treatment that provides patients with adequate hydration and nutrition. However, NG is easily dislodged after a long duration of placement; furthermore, lacking accurate feeding skills could also lead to aspiration pneumonia.

DETAILED DESCRIPTION:
Aspiration pneumonia is a common complication in senior patients with high morbidity and mortality rate. The decline of physical function among elders can easily lead to swallowing disorders, and nasogastric (NG) tube insertion is an emergency medical treatment that provides patients with adequate hydration and nutrition. However, NG is easily dislodged after a long duration of placement; furthermore, lacking accurate feeding skills could also lead to aspiration pneumonia. An appropriate NG care model to lower feeding complications is an essential issue. The purpose of this study is to investigate the efficacy of eating rehabilitation training in the removal of NG tubes among elderly patients with aspiration pneumonia. This is an experimental, convenient sampling study. We enrolled first-time NG tube insertion friends and complicated with aspiration pneumonia. All patients in this study were from the medical ward of a tertiary center in northern Taiwan. The target numbers are ninety-six patients. The eligible subjects will be randomized to the experimental and the control group. The experimental group will receive eating rehabilitation training, including oral care, saliva gland massage, oral exercise, feeding strategy, and swallowing skill education. The control group will receive routine medical care. The endpoint of this study includes 1. The timing of NG removal, 2. The re-insertion rate after one month of NG removal, 3. 30 days unexpected re-admission rate. The characteristics and distribution of variables were described by percentage, mean, and standard deviation. The Chi-square test was used to analyze the difference between-group differences on the 30 days of NG re-insertion and re-admission rate. The timing of NG removal between the two groups was analyzed by Kaplan-Meier survival. All statistical analyses were performed on Statistical Package for Social Sciences (SPSS) version 22.0. This study's results provide caregivers with more successful strategy for removing senior aspiration pneumonia patients' nasogastric tubes and improving early oral intake and patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients than or equal to 75 years old
2. Clear consciousness
3. Diagnosed with aspiration pneumonia (the main diagnostic disease code is ICD-9-CM: 507; ICD-10-CM: J69)
4. Those who were hospitalized for more than 24 hours and had a nasogastric tube inserted for the first time within 1 month
5. Those who can communicate in Chinese or Taiwanese
6. The doctor judges that the condition is stable, such as: body temperature < 37.5°C, heart rate < 100 beats/min, respiratory rate < 24/min, systolic blood pressure > 90 mmHg and fingertip pulse oximeter saturation greater than 90%

Exclusion Criteria:

1. Patients who have been placed in a nasogastric tube or gastrostomy for force-feeding before seeing a doctor
2. Diagnosed with other neurological disorders, such as Parkinson's disease, multiple sclerosis, polio, dermatomyosclerosis inflammation, and myasthenia gravis
3. Those who use oxygen masks or respirators

Ages: 75 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
nasogastric tube successfully removed and spent of time with removed successfully nasogastric tube | From date of randomization until the date of discharge from the cause, assessed up to one month.
  It was observed from the bedside that the subjects had successfully removed the nasogastric tube according to the doctor's advice before being discharged from the hospital. The criteria for successfully removing the nasogastric tube in the ward include: the research subject can accept oral medication, can eat about 1000ml per day, and has no cough when eating. In addition to the above circumstances, when removing the nasogastric tube, the doctor's confirmation and removal of the doctor's order are also required

SECONDARY OUTCOMES:
The re-insertion rate after one month of NG removal | From the date of discharge from any cause, assessed up to one month.
  Subjects whose nasogastric tube was removed during hospitalization were followed up at the bedside or by telephone once a week after the removal of the nasogastric tube to find out whether there was any unexpected nasogastric tube re-insertion within 30 days after the removal of the nasogastric tube.

OTHER OUTCOMES:
30 days unexpected re-admission rate. | From the date of discharge from any cause, assessed up to one month.
  It refers to the rate of rehospitalization due to pneumonia on the 30th day from the date of discharge for patients who are unexpectedly readmitted within the 30th day from the date of discharge from the medical records of each research subject.

CONTACTS AND LOCATIONS:
Overall Officials: Tase Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen S, Kent B, Cui Y. Interventions to prevent aspiration in older adults with dysphagia living in nursing homes: a scoping review. BMC Geriatr. 2021 Jul 17;21(1):429. doi: 10.1186/s12877-021-02366-9. PMID 34273953
- [Background] Averin A, Shaff M, Weycker D, Lonshteyn A, Sato R, Pelton SI. Mortality and readmission in the year following hospitalization for pneumonia among US adults. Respir Med. 2021 Aug-Sep;185:106476. doi: 10.1016/j.rmed.2021.106476. Epub 2021 May 21. PMID 34087608
- [Background] Baijens LW, Clave P, Cras P, Ekberg O, Forster A, Kolb GF, Leners JC, Masiero S, Mateos-Nozal J, Ortega O, Smithard DG, Speyer R, Walshe M. European Society for Swallowing Disorders - European Union Geriatric Medicine Society white paper: oropharyngeal dysphagia as a geriatric syndrome. Clin Interv Aging. 2016 Oct 7;11:1403-1428. doi: 10.2147/CIA.S107750. eCollection 2016. PMID 27785002
- [Background] Chauhan D, Varma S, Dani M, Fertleman MB, Koizia LJ. Nasogastric Tube Feeding in Older Patients: A Review of Current Practice and Challenges Faced. Curr Gerontol Geriatr Res. 2021 Jan 21;2021:6650675. doi: 10.1155/2021/6650675. eCollection 2021. PMID 33936197
- [Background] Chen HH, Lin PY, Lin CK, Lin PY, Chi LY. Effects of oral exercise on tongue pressure in Taiwanese older adults in community day care centers. J Dent Sci. 2022 Jan;17(1):338-344. doi: 10.1016/j.jds.2021.10.017. Epub 2021 Nov 27. PMID 35028056